CLINICAL TRIAL: NCT03569709
Title: Guided Aerobic Exercise Therapy to Improve Recovery From Acute Concussion: A Randomized Controlled Trial
Brief Title: Early Sub-threshold Exercise Treatment for Concussion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Harvard University (Other); The Mind Research Network (Other)
Responsible Party: Principal Investigator, John J. Leddy MD, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1 R01 NS106260-01
Record Dates: First submitted 2018-06-05; First posted 2018-06-26 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Active Comparator): Sub-threshold aerobic exercise.
  Interventions: Behavioral: Aerobic Exercise
- Stretching (Placebo Comparator): Stretching program that will not raise heart rate.
  Interventions: Behavioral: Stretching
- Rest (Placebo Comparator): Relative rest. Avoid all structured exercise.
  Interventions: Behavioral: Rest

INTERVENTIONS:
Behavioral: Aerobic Exercise — Progressive sub-threshold aerobic exercise
  Arms: Aerobic Exercise
Behavioral: Rest — No structured exercise.
  Arms: Rest
Behavioral: Stretching — Gentle progressive upper and lower extremity stretching program
  Arms: Stretching

SUMMARY:
Each year millions of Americans suffer concussions as a result of accidents in sports, at work or through military service. Adolescents take the longest to recover from the effects of concussion yet no therapy exists to help speed their recovery. This project aims to see if a program of early guided aerobic exercise can safely speed recovery from concussion in adolescents and investigates some reasons for why this type of therapy could be effective.

DETAILED DESCRIPTION:
Most children with concussion recover spontaneously within 2-4 weeks of injury but approximately 30% experience prolonged post-concussive symptoms (PPCS), impacting quality of life. There are no evidence-based therapies for acute pediatric concussion. Instead, current consensus-based-recommendations include physical and cognitive rest as the mainstays of treatment despite evidence to the contrary that excessive rest prolongs recovery and that early (first week) activity reduces PPCS incidence. The investigators were the first to demonstrate that a systematic evaluation of exercise tolerance using the Buffalo Concussion Treadmill Test (BCTT) to prescribe a guided exercise prescription in those with PPCS safely sped recovery. The investigators have preliminary data that exercise may speed recovery if administered within the first week after sport-related concussion (SRC). Concussion is associated with adverse effects on the autonomic nervous system (ANS) and control of cerebral blood flow (CBF). The investigators have shown that sub-threshold aerobic exercise reduces symptoms in PPCS in association with normalization of ANS function and CBF control, providing a potential mechanism of action as well as target engagement for this non-pharmacological therapy. An important translational aspect is that the BCTT would be for clinicians a clinical proxy of concussion physiology that would help make the difficult return-to-activity/play decision more objective and physiologically-based. The investigators' long-term goals are to develop therapies that safely speed recovery from concussion, return youth back to their typical activities, actively prevent PPCS, and develop practical physiological tools for clinicians. The overall objective of this application is to determine if early guided aerobic exercise speeds recovery from SRC. The investigators specifically test underlying mechanisms of action for faster recovery by measuring ANS function (the cold pressor test, CPT) and CBF (by Arterial Spin Labeling, ASL). Age- and sex-matched healthy controls will be recruited to quantify physiological CBF differences and serve as a normative control group. The investigators will examine these questions in a randomized, multisite controlled trial in adolescents aged 13-18y with acute SRC by pursuing the following two specific aims: (1) determine if guided aerobic exercise/education speeds recovery after acute concussion in adolescents compared with (a) rest/education with a gradual return to activities, (i.e., current recommendation) and (b) a progressive stretching program/education (attention placebo); and (2) as secondary aims the investigators will quantify the effects of each intervention in Aim 1 on CBF and on autonomic function (CPT), which serve as relevant and objective physiological measures of autonomic regulation of CBF following concussion. This project will provide critical evidence to support the role of guided aerobic exercise for the active treatment of acute concussion and for a physiological mechanism(s) for its effect, which would lead to a paradigm shift from the current passive approach to treatment. The translational aspect of the project is unique and would have immediate impact to help clinicians determine recovery based on physiology rather than symptoms. A controlled active approach to concussion treatment may also substantially reduce the incidence of PPCS in children.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years; any race, ethnicity, or sex.
* Concussion sustained 2-7 days prior to first clinical visit.
* Symptom score (new symptoms) >3 on the Post-Concussion Symptom Inventory Scale.
* Glasgow Coma Scale (GCS) of 13-15 (if available in medical record), an alteration in mental status, loss of consciousness (if present) of less than 30 minutes, and post-traumatic amnesia (if present) limited to <24 hours.
* Low risk for cardiac disease and willing to exercise.
* Medications, except for βeta- and calcium-blockers, are acceptable.

Exclusion Criteria:

* GCS score <13 at time of injury.
* Lesion on CT/MRI (via review of emergency department records) and/or focal neurologic deficit consistent with an intracerebral lesion (e.g., unilateral weakness, dilated pupil).
* Inability to exercise because of orthopedic injury, significant vestibular dysfunction, visual abnormality, or increased cardiac risk.
* Neurosurgical intervention, general anesthesia and previously diagnosed neurological or psychiatric diseases.
* Additional head injury after study enrollment.
* Active substance abuse/dependence.
* Non-fluency in English.
* βeta- and calcium blocker use.
* Autism, metal braces or other metal that would interfere with ASL.
* Unwilling to exercise.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | up to 2 days
  Time to baseline level of symptoms on Post Concussion Symptom Inventory (PCSI) for 2 days in a row

SECONDARY OUTCOMES:
Autonomic function | Within one week of injury and at 1 month after injury
  Autonomic function as assessed by the Cold Pressor Test (CPT)
Delayed recovery | 1 and 4 months after concussion
  Persistence of increased symptoms on the PCSI at 1 and at 4 months after concussion
Cerebral Blood Flow (CBF) | Within one week of injury and at 1 month after injury
  CBF by Arterial Spin Labelling MRI

IPD SHARING:
Plan to Share IPD: No